CLINICAL TRIAL: NCT04901130
Title: Impact of Real-time Automatic Quality Control System on Colorectal Adenoma Detection: a Multicenter Randomized Controlled Trial
Brief Title: Impact of Real-time Automatic Quality Control System on Colorectal Adenoma Detection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Collaborators: Binzhou Medical University (Other); Shengli Oilfield Hospital (Other); Linyi People's Hospital (Other); Zibo Municipal Hospital (Other); The People's Hospital of Zhaoyuan City (Unknown)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2021SDU-QILU-066
Record Dates: First submitted 2021-05-24; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Colonoscopy
Keywords: Artificial Intelligence; Colonoscopy; Quality Control

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AQCS-aided group (Experimental): Patients in AQCS-aided group will go through colonoscopy examination with the assitance of AQCS.
  Interventions: Device: Computer-aided Real-time Automatic Quality Control System (AQCS)
- Control group (No Intervention): Patients in control group will go through conventional standard colonoscopy examination without the assistance of the AQCS.

INTERVENTIONS:
Device: Computer-aided Real-time Automatic Quality Control System (AQCS) — Automatic quality-control system(AQCS), developed based on deep convolutional neural network (DCNN) models, could improve the colonoscopists' performance during withdrawal phase and significantly increase polyp and adenoma detection.
  Arms: AQCS-aided group

SUMMARY:
The purpose of this study was to assess the performance of automatic quality-control system (AQCS) in real-time quality control of colonoscopy.

DETAILED DESCRIPTION:
We carried a multicenter randomised controlled trial to assess the performance of this system in quality control of real-time colonoscopy, including the adenoma detection rate (ADR), withdraw time, adequate bowel preparation rate and other indicators.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients (aged 18-80 years) scheduled for colonoscopy examination.

Exclusion Criteria:

* Patients with a history of inflammatory bowel disease, advanced colorectal cancer, polyposis syndromes or known colorectal polyps without complete removal previously.
* Patients with a history of colorectal surgery.
* Patients with a contraindication for biopsy.
* Patients with prior failed colonoscopy.
* Patients with known stenosis or obstruction.
* Patients in pregnancy or lactation phase.
* Patients refused to participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1254 (Estimated)
Dates: Start 2021-05-27 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Colorectal adenoma detection rate (ADR) | 10 months
  The primary endpoint is the adenoma detection rate (ADR), which is the proportion of patients having one or more adenomas detected by colonoscopy.

SECONDARY OUTCOMES:
Colorectal polyp detection rate (PDR) | 10 months
  The polyp detection rate (PDR) is the proportion of patients having one or more polyps detected by colonoscopy.
The mean number of adenomas detected per colonoscopy (APC) | 10 months
  The mean number of adenomas detected per colonoscopy in AQCS and control groups
The mean number of polyps detected per colonoscopy (PPC) | 10months
  The mean number of polyps detected per colonoscopy in AQCS and control groups
Withdrawl time | During procedure
  Withdrawl time is defined as the time taken to remove the colonoscope from the cecal pole minus the time of therapeutic interventions or biopsy, until the complete withdrawal of the colonoscope.

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD, Study Chair — Qilu Hospital of Shandong University; Xiuli Zuo, PhD, Study Chair — Qilu Hospital of Shandong University
Locations (6):
- China (6):
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Linyi People's Hospital, Dezhou, Shandong
  - Central Hospital of Shengli Oilfield, Dongying, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The People's Hospital of Zhaoyuan City, Yantai, Shandong
  - Zibo Municipal Hospital, Zibo, Shandong

REFERENCES:
- [Derived] Liu J, Zhou R, Liu C, Liu H, Cui Z, Guo Z, Zhao W, Zhong X, Zhang X, Li J, Wang S, Xing L, Zhao Y, Ma R, Ni J, Li Z, Li Y, Zuo X. Automatic Quality Control System and Adenoma Detection Rates During Routine Colonoscopy: A Randomized Clinical Trial. JAMA Netw Open. 2025 Jan 2;8(1):e2457241. doi: 10.1001/jamanetworkopen.2024.57241. PMID 39883463